CLINICAL TRIAL: NCT02269917
Title: A Phase 3, Randomized, Active-controlled, Open-label Study to Evaluate the Efficacy, Safety and Tolerability of Switching to a Darunavir/ Cobicistat/ Emtricitabine/ Tenofovir Alafenamide (D/C/F/TAF) Once-daily Single-tablet Regimen Versus Continuing the Current Regimen Consisting of a Boosted Protease Inhibitor (bPI) Combined With Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF) in Virologically-suppressed, Human Immunodeficiency Virus Type 1 (HIV-1) Infected Subjects
Brief Title: Study to Evaluate Efficacy and Safety of Darunavir/Cobicistat/Emtricitabine/Tenofovir Alafenamide (D/C/F/TAF) Regimen Versus Boosted Protease Inhibitor (bPI) Along With Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF) Regimen in Virologically-Suppressed, HIV-1 Infected Participants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen R&D Ireland (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR105736; TMC114IFD3013 (Other: Janssen R&D Ireland); 2014-003052-31 (EudraCT Number)
Record Dates: First submitted 2014-10-17; First posted 2014-10-21 (Estimated); Results first posted 2018-11-09 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-11

CONDITIONS: Human Immunodeficiency Virus Type 1
Keywords: Human Immunodeficiency Virus Type 1; Emerald; Darunavir; Cobicistat; Emtricitabine; Tenofovir Alafenamide
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental Treatment Regimen (Experimental): Participants will receive a single fixed dose combination (FDC) tablet containing darunavir (DRV) 800 milligram (mg)/ cobicistat (COBI) 150 mg/ emtricitabine (FTC) 200 mg/ tenofovir alafenamide (TAF) 10 mg (D/C/F/TAF tablet), orally once daily, up to Week 48. After Week 48, all participants will continue to receive the D/C/F/TAF tablet in a 48 week extension phase (up to Week 96).
  Interventions: Drug: D/C/F/TAF
- Current Treatment Regimen (Active Comparator): Participants will receive a boosted protease inhibitor (bPI) (limited to darunavir [DRV] or atazanavir with low-dose ritonavir [rtv] or cobicistat [COBI], or lopinavir with rtv) combined with emtricitabine/tenofovir disoproxil fumarate (FTC/TDF) up to Week 52. After Week 52, all participants will receive the D/C/F/TAF tablet in a 44 week extension phase (up to Week 96).
  Interventions: Drug: Boosted Protease Inhibitor (bPI); Drug: FTC/TDF

INTERVENTIONS:
Drug: D/C/F/TAF — Once-daily single-tablet regimen containing darunavir (DRV) 800 milligram (mg)/ cobicistat (COBI) 150 mg/ emtricitabine (FTC) 200 mg/ tenofovir alafenamide (TAF) 10 mg.
  Arms: Experimental Treatment Regimen
Drug: Boosted Protease Inhibitor (bPI) — Boosted protease inhibitor (limited to darunavir [DRV] or atazanavir with low-dose ritonavir [rtv] or cobicistat [COBI], or lopinavir with rtv) as per current treatment regimen.
  Arms: Current Treatment Regimen
Drug: FTC/TDF — Emtricitabine/tenofovir disoproxil fumarate (FTC/TDF).
  Arms: Current Treatment Regimen

SUMMARY:
The purpose of this study is to demonstrate non-inferiority in efficacy while switching to a once-daily single-tablet regimen containing darunavir (DRV)/ cobicistat (COBI)/ emtricitabine (FTC)/ tenofovir alafenamide (TAF) (D/C/F/TAF tablet) relative to continuing the current regimen consisting of a boosted protease inhibitor (bPI) combined with tenofovir disoproxil fumarate (FTC/TDF) in virologically-suppressed (human immunodeficiency virus type 1 ribonucleic acid [HIV-1 RNA] concentrations less than [<] 50 copies per milliliter [copies/mL]) HIV-1 infected participants.

DETAILED DESCRIPTION:
This is a randomized (study medication assigned to participants by chance), active-controlled (study in which the experimental treatment or procedure is compared to a standard treatment or procedure), open-label (participants and researchers are aware about the treatment, participants are receiving), multicenter (when more than 1 hospital or medical school team work on a medical research study), study in virologically-suppressed, HIV-1 infected adult participants. The study will include a Screening Period of approximately 30 days (up to maximum 6 weeks), a controlled Treatment Period of 48 weeks, an Extension Phase of 48 weeks. All eligible participants will be randomly assigned to receive either current treatment regimen - a bPI (limited to DRV with low-dose ritonavir [rtv] or COBI, atazanavir [ATV] with rtv or COBI, or lopinavir [LPV] with rtv) combined with FTC/TDF, or experimental treatment regimen - D/C/F/TAF once-daily single-tablet for 48 weeks. After completion of week 48, participants assigned to the experimental treatment will continue with D/C/F/TAF in the extension phase up to week 96 . Participants who continued their current regimen will receive the experimental treatment (if all criteria are fulfilled) at week 52 up to week 96. As from Week 96, all participants will be given the option to continue D/C/F/TAF treatment, if they wish and if they continue to benefit from it until D/C/F/TAF becomes commercially available and is reimbursed, or can be accessed through another source in the country where he/she is living,or until the sponsor terminates clinical development. A bone investigation substudy will be performed at selected study sites, to assess bone biomarkers and energy x-ray absorptiometry (DXA) scans, in approximately 300 participants (200 in the D/C/F/TAF treatment arm versus 100 in the control arm) who provide informed consent for the substudy.

ELIGIBILITY:
Inclusion Criteria:

* Currently being treated with a stable antiretroviral (ARV) regimen consisting of a boosted protease inhibitor (limited to darunavir [DRV] or atazanavir with low-dose ritonavir [rtv] or cobicistat [COBI], or lopinavir with rtv) combined with emtricitabine/tenofovir disoproxil fumarate (FTC/TDF) only, for at least 6 consecutive months preceding the Screening visit
* On-treatment plasma human immunodeficiency virus type 1 ribonucleic acid (HIV-1 RNA) concentrations less than (<) 50 copies per milliliter (copies/mL) or HIV-1 RNA undetectable by a local HIV-1 RNA test between 12 and 2 months prior to the Screening visit and have HIV-1 RNA <50 copies/mL at the Screening visit
* A single virologic elevation of greater than or equal to (>=) 50 copies/mL after previously reaching viral suppression between 12 and 2 months prior to Screening is acceptable, provided a subsequent test prior to Screening was <50 copies/mL
* Absence of history of failure on DRV treatment and absence of DRV resistance-associated mutations (RAMs), if documented historical genotypes are available
* Normal electrocardiogram (ECG) at Screening (or if abnormal, determined by the Investigator to be not clinically significant)

Exclusion Criteria:

* A new acquired immunodeficiency syndrome (AIDS) - defining condition diagnosed within the 30 days prior to Screening
* Proven or suspected acute hepatitis within 30 days prior to study entry
* Hepatitis C antibody positive; however, participants previously cured of hepatitis C virus (HCV) infection, with documented sustained virologic response, that is, undetectable HCV RNA 24 weeks after the last dose of HCV treatment, are allowed to participate
* Hepatitis B surface antigen (HBsAg) positive
* Participants with cirrhosis as diagnosed based on local practices

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1149 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2020-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen R&D Ireland Clinical Trial, Study Director — Janssen R&D Ireland
Locations (79):
- United States (38):
  - Phoenix, Arizona
  - Bakersfield, California
  - Beverly Hills, California
  - Long Beach, California
  - Los Angeles, California
  - San Diego, California
  - San Francisco, California
  - Washington D.C., District of Columbia
  - Fort Lauderdale, Florida
  - Ft. Pierce, Florida
  - Orlando, Florida
  - West Palm Beach, Florida
  - Atlanta, Georgia
  - Savannah, Georgia
  - Chicago, Illinois
  - Boston, Massachusetts
  - Springfield, Massachusetts
  - Berkley, Michigan
  - Detroit, Michigan
  - Minneapolis, Minnesota
  - Kansas City, Missouri
  - St Louis, Missouri
  - Hillsborough, New Jersey
  - Newark, New Jersey
  - Somers Point, New Jersey
  - Santa Fe, New Mexico
  - New York, New York
  - Chapel Hill, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Philadelphia, Pennsylvania
  - Providence, Rhode Island
  - Austin, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Longview, Texas
  - Seattle, Washington
- Belgium (5):
  - Antwerp
  - Brussels
  - Ghent
  - Leuven
  - Liège
- Canada (4):
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Toronto, Ontario
  - Montreal, Quebec
- France (8):
  - Le Kremlin-Bicêtre
  - Lyon
  - Marseille
  - Montpellier
  - Nantes
  - Paris
  - Strasbourg
  - Tourcoing
- Poland (5):
  - Bydgoszcz
  - Chorzów
  - Lodz
  - Warsaw
  - Wroclaw
- San Juan, Puerto Rico
- Spain (9):
  - Alicante
  - Badalona
  - Barcelona
  - Córdoba
  - Donostia / San Sebastian
  - Elche
  - Madrid
  - Seville
  - Valencia
- Sweden (3):
  - Gothenburg
  - Malmo
  - Stockholm
- Switzerland (3):
  - Basel
  - Bern
  - Zurich
- United Kingdom (3):
  - Brighton
  - London
  - Manchester

REFERENCES:
- [Derived] Ackaert O, McDougall D, Perez-Ruixo C, Perez-Ruixo JJ, Jezorwski J, Crauwels HM. Population Pharmacokinetic Analysis of Darunavir and Tenofovir Alafenamide in HIV-1-Infected Patients on the Darunavir/Cobicistat/Emtricitabine/Tenofovir Alafenamide Single-Tablet Regimen (AMBER and EMERALD Studies). AAPS J. 2021 Jun 7;23(4):82. doi: 10.1208/s12248-021-00607-8. PMID 34100149
- [Derived] Huhn GD, Wilkin A, Mussini C, Spinner CD, Jezorwski J, El Ghazi M, Van Landuyt E, Lathouwers E, Brown K, Baugh B; AMBER and EMERALD study groups. Week 96 subgroup analyses of the phase 3, randomized AMBER and EMERALD trials evaluating the efficacy and safety of the once daily darunavir/cobicistat/emtricitabine/tenofovir alafenamide (D/C/F/TAF) single-tablet regimen in antiretroviral treatment (ART)-naive and -experienced, virologically-suppressed adults living with HIV-1. HIV Res Clin Pract. 2020 Dec;21(6):151-167. doi: 10.1080/25787489.2020.1844520. Epub 2021 Feb 2. PMID 33528318
- [Derived] Lathouwers E, Wong EY, Brown K, Baugh B, Ghys A, Jezorwski J, Mohsine EG, Van Landuyt E, Opsomer M, De Meyer S; AMBER and EMERALD Study Groups. Week 48 Resistance Analyses of the Once-Daily, Single-Tablet Regimen Darunavir/Cobicistat/Emtricitabine/Tenofovir Alafenamide (D/C/F/TAF) in Adults Living with HIV-1 from the Phase III Randomized AMBER and EMERALD Trials. AIDS Res Hum Retroviruses. 2020 Jan;36(1):48-57. doi: 10.1089/AID.2019.0111. Epub 2019 Oct 21. PMID 31516033
- [Derived] Huhn GD, Eron JJ, Girard PM, Orkin C, Molina JM, DeJesus E, Petrovic R, Luo D, Van Landuyt E, Lathouwers E, Nettles RE, Brown K, Wong EY. Darunavir/cobicistat/emtricitabine/tenofovir alafenamide in treatment-experienced, virologically suppressed patients with HIV-1: subgroup analyses of the phase 3 EMERALD study. AIDS Res Ther. 2019 Aug 29;16(1):23. doi: 10.1186/s12981-019-0235-1. PMID 31464642
- [Derived] Orkin C, Molina JM, Negredo E, Arribas JR, Gathe J, Eron JJ, Van Landuyt E, Lathouwers E, Hufkens V, Petrovic R, Vanveggel S, Opsomer M; EMERALD study group. Efficacy and safety of switching from boosted protease inhibitors plus emtricitabine and tenofovir disoproxil fumarate regimens to single-tablet darunavir, cobicistat, emtricitabine, and tenofovir alafenamide at 48 weeks in adults with virologically suppressed HIV-1 (EMERALD): a phase 3, randomised, non-inferiority trial. Lancet HIV. 2018 Jan;5(1):e23-e34. doi: 10.1016/S2352-3018(17)30179-0. Epub 2017 Oct 6. PMID 28993180

RESULTS

PARTICIPANT FLOW:
Groups:
- D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]): Participants received a single fixed dose combination (FDC) tablet containing darunavir (DRV) 800 milligram (mg)/ cobicistat (COBI) 150 mg/ emtricitabine (FTC) 200 mg/ tenofovir alafenamide (TAF) 10 mg (D/C/F/TAF tablet), orally once daily up to Week 48. After Week 48, all participants continued to receive D/C/F/TAF treatment (that is, initial switch to D/C/F/TAF group) up to Week 96. After Week 96, participants were given the opportunity to continue D/C/F/TAF treatment until D/C/F/TAF became commercially available up to 42 months (end of extension).
- Control (Baseline to Switch): Participants received a boosted protease inhibitor (bPI) (limited to darunavir [DRV] or atazanavir with low-dose ritonavir [rtv] or cobicistat [COBI], or lopinavir with rtv) combined with emtricitabine/tenofovir disoproxil fumarate (F/TDF) up to Week 48.
- Switch to D/C/F/TAF: After Week 52, participants earlier receiving treatment with bPI+F/TDF switched to D/C/F/TAF treatment up to Week 96. After Week 96, participants were given the opportunity to continue D/C/F/TAF treatment until D/C/F/TAF became commercially available for up to 42 months.
Period: BL to EOE-Test and BL to Switch-Control
Arm/Group | D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) | Control (Baseline to Switch) | Switch to D/C/F/TAF
Started | 766 | 383 | 0
Treated | 763 | 378 | 0
Completed | 649 | 352 | 0
Not Completed | 117 | 31 | 0
Not completed — Lost to Follow-up | 25 | 7 | 0
Not completed — Other | 19 | 4 | 0
Not completed — Withdrawal by Subject | 32 | 10 | 0
Not completed — Adverse Event | 24 | 4 | 0
Not completed — Non-compliance with study drug | 4 | 0 | 0
Not completed — Physician Decision | 4 | 0 | 0
Not completed — Protocol Violation | 2 | 1 | 0
Not completed — Death | 4 | 0 | 0
Not completed — Randomized but not treated | 3 | 5 | 0
Period: Switch to D/C/F/TAF (Until EOE)
Arm/Group | D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) | Control (Baseline to Switch) | Switch to D/C/F/TAF
Started | 0 | 0 | 352
Completed | 0 | 0 | 314
Not Completed | 0 | 0 | 38
Not completed — Death | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 10
Not completed — Adverse Event | 0 | 0 | 11
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Pregnancy | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 5
Not completed — Other | 0 | 0 | 8

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) analysis set included all the participants who were randomized and received at least 1 dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) | Control (Baseline to Switch) | Total
Number analyzed (Participants) | 763 | 378 | 1141
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.3 (10.86) | 44.8 (10.77) | 45.1 (10.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 140 | 65 | 205
  Male | 623 | 313 | 936
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 111 | 59 | 170
  Not Hispanic or Latino | 649 | 317 | 966
  Unknown or Not Reported | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 2 | 7
  Asian | 17 | 9 | 26
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 155 | 82 | 237
  White | 573 | 282 | 855
  More than one race | 5 | 1 | 6
  Unknown or Not Reported | 6 | 2 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 17 | 9 | 26
  Black or African American | 155 | 82 | 237
  Hispanic or Latino | 95 | 56 | 151
  Other | 20 | 6 | 26
  White Non-Hispanic | 476 | 225 | 701
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 32 | 20 | 52
  Canada | 45 | 21 | 66
  France | 69 | 28 | 97
  Poland | 91 | 35 | 126
  Spain | 117 | 52 | 169
  Sweden | 23 | 5 | 28
  Switzerland | 26 | 13 | 39
  United Kingdom | 47 | 23 | 70
  United States | 313 | 181 | 494

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Virologic Rebound (HIV-1 RNA >=50 Copies/mL) Cumulative Through Week 48
Description: Virologic rebound was defined as: confirmed plasma human immunodeficiency virus - 1 (HIV-1) Ribonucleic Acid (RNA) level greater than or equal to (>=)50 copies per milliliter (copies/mL) up to, and including the upper bound of the Week 48 window (ie, 54 weeks) and last available on-treatment (single) HIV-1 RNA >=50 copies/mL at premature discontinuation (irrespective of reason). Percentage of participants with virologic rebound were reported.
Time Frame: Through Week 48
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) | Control (Baseline to Switch)
Number analyzed (Participants) | 763 | 378
Percentage of participants | 2.5 [1.5 to 3.9] | 2.1 [0.9 to 4.1]
Statistical Analysis 1: Comparison: D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) vs Control (Baseline to Switch); Test type: Non-Inferiority — 4; p < 0.001, Stratum-adjusted Mantel-Haenszel (MH); Difference in percentage = 0.4, 95% CI 2-sided [-1.5 to 2.2]

2. Secondary Outcome: Percentage of Participants With Virologic Rebound (Plasma HIV-1 RNA >=20 Copies/mL) Cumulative Through 48 Weeks
Description: Virologic rebound was defined as: confirmed plasma HIV-1 RNA >=20 copies/mL up to, and including the upper bound of the Week 48 window (ie, 54 weeks) and last available on-treatment (single) HIV-1 RNA >=20 copies/mL at premature discontinuation (irrespective of reason). Percentage of participants with virologic rebound were reported.
Time Frame: Through 48 Weeks
Population: ITT analysis set included all participants who were randomized and received at least 1 dose of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) | Control (Baseline to Switch)
Number analyzed (Participants) | 763 | 378
Percentage of Participants | 10.5 [8.4 to 12.9] | 11.4 [8.4 to 15.0]

3. Secondary Outcome: Percentage of Participants With Virologic Rebound (Plasma HIV-1 RNA >=200 Copies/mL) Cumulative Through 48 Weeks
Description: Virologic rebound was defined as: confirmed plasma HIV-1 RNA >=200 copies/mL up to, and including the upper bound of the Week 48 window (ie, 54 weeks) and last available on-treatment (single) HIV-1 RNA >=200 copies/mL at premature discontinuation (irrespective of reason). Percentage of participants with virologic rebound were reported.
Time Frame: Through 48 Weeks
Population: ITT analysis set included all participants who were randomized and received at least 1 dose of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) | Control (Baseline to Switch)
Number analyzed (Participants) | 763 | 378
Percentage of Participants | 0.4 [0.1 to 1.1] | 0.0 [NA to NA] — Here NA signifies that the Confidence Interval (CI) was not estimable as no participants had virologic rebound in this group.

4. Secondary Outcome: Percentage of Participants With Non-Virologic Rebound at Week 48 by Kaplan-Meier Estimates
Description: Virologic rebound was defined as: confirmed plasma HIV-1 RNA >=50 copies/mL up to, and including the upper bound of the Week 48 window (ie, 54 weeks) and last available on-treatment (single) HIV-1 RNA >=50 copies/mL at premature discontinuation (irrespective of reason). Here Kaplan-Meier estimates percentage of participants with non-virologic rebound at week 48.
Time Frame: Baseline up to Week 48
Population: ITT analysis set included all participants who were randomized and received at least 1 dose of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) | Control (Baseline to Switch)
Number analyzed (Participants) | 763 | 378
percentage of participants | 97.7 [96.4 to 98.6] | 97.8 [95.7 to 98.9]

5. Secondary Outcome: Percentage of Participants Experiencing Grade 3 and 4 Adverse Events (AEs), Serious Adverse Events (SAEs), and Premature Discontinuation Due to AEs Through Week 48
Description: An AE is any untoward medical occurrence in participant who received study drug without regard to possibility of causal relationship. Grade 3 (Severe) events were symptoms causing inability to perform usual social & functional activities. Grade 4 (Life-threatening) events were symptoms causing inability to perform basic self-care functions or medical or operative intervention indicated to prevent permanent impairment, persistent disability, or death.
Time Frame: Up to Week 48
Population: ITT analysis set included all the participants who were randomized and received at least 1 dose of study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) | Control (Baseline to Switch)
Number analyzed (Participants) | 763 | 378
Percentage of Participants
  Grade 3 AEs | 5.6 | 6.3
  Grade 4 AEs | 1.2 | 1.9
  SAEs | 4.6 | 4.8
  Premature discontinuations due to AEs | 1.4 | 1.3

6. Secondary Outcome: Change From Baseline in Serum Creatinine Levels at Weeks 24 and 48
Description: Change from baseline in serum creatinine levels at Weeks 24 and 48 was assessed.
Time Frame: Baseline and Weeks 24 and 48
Population: ITT analysis set included all participants randomized and received at least 1 dose of study treatment. Here, N (number of participants analyzed) indicates number of participants evaluable for this endpoint; and 'n' specifies participants analyzed for this endpoint at given time point.
Measure: Least Squares Mean (Standard Error); unit: micro mole per liter
Arm/Group | D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) | Control (Baseline to Switch)
Number analyzed (Participants) | 761 | 378
micro mole per liter
  Change at Week 24: number analyzed (Participants) | 735 | 362
  Change at Week 24 | 1.22 (0.358) | 0.88 (0.509)
  Change at Week 48: number analyzed (Participants) | 725 | 350
  Change at Week 48 | 1.27 (0.368) | 0.65 (0.530)
Statistical Analysis 1: Comparison: D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) vs Control (Baseline to Switch); Change at Week 24; Test type: Other; p = 0.580, ANCOVA; Least Square (LS) Mean Difference = 0.34, 95% CI 2-sided [-0.88 to 1.57], Standard Error of Mean 0.623
Statistical Analysis 2: Comparison: D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) vs Control (Baseline to Switch); Change at Week 48; Test type: Other; p = 0.340, ANCOVA; Least Square (LS) Mean Difference = 0.62, 95% CI 2-sided [-0.65 to 1.88], Standard Error of Mean 0.646

7. Secondary Outcome: Change From Baseline in Estimated Glomerular Filtration Rate Based on Serum Creatinine (eGFRcr, by Cockcroft-Gault Formula [eGFRcg]) at Weeks 24 and 48
Description: Change from baseline in eGFRcr (by Cockcroft-Gault formula) was assessed at Weeks 24 and 48. eGFRcr according to the Cockcroft Gault formula- Male: (140 - age in years)*(weight in kilogram [kg])/72*(serum creatinine in milligram per deciliter [mg/dL])=eGFRcr (milliliter per minute [mL/min]); Female: (140 - age in years)*(weight in kg)/72*(serum creatinine in mg/dL)*0.85=eGFRcr (mL/min).
Time Frame: Baseline, Weeks 24 and 48
Population: ITT analysis set included all the participants who were randomized and received at least 1 dose of study treatment. Here, N (number of participants analyzed) indicates number of participants evaluable for this endpoint; and 'n' specifies those participants who were analyzed for this endpoint at given time point.
Measure: Least Squares Mean (Standard Error); unit: milliliter per minute (mL/min)
Arm/Group | D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) | Control (Baseline to Switch)
Number analyzed (Participants) | 761 | 378
milliliter per minute (mL/min)
  Change at Week 24: number analyzed (Participants) | 735 | 362
  Change at Week 24 | -0.38 (0.502) | 0.20 (0.715)
  Change at Week 48: number analyzed (Participants) | 725 | 350
  Change at Week 48 | -0.94 (0.492) | -0.20 (0.708)
Statistical Analysis 1: Comparison: D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) vs Control (Baseline to Switch); Change at Week 24; Test type: Other; p = 0.506, ANCOVA; LS Mean Difference = -0.58, 95% CI 2-sided [-2.30 to 1.13], Standard Error of Mean 0.874
Statistical Analysis 2: Comparison: D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) vs Control (Baseline to Switch); Change Week 48; Test type: Other; p = 0.392, ANCOVA; LS Mean Difference = -0.74, 95% CI 2-sided [-2.43 to 0.95], Standard Error of Mean 0.862

8. Secondary Outcome: Change From Baseline in Estimated Glomerular Filtration Rate Based on Serum Creatinine (eGFRcr, by Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI]) at Weeks 24 and 48
Description: Change from baseline in eGFRcr (by CKD-EPI) was assessed at Weeks 24 and 48. eGFRcr per CKD-EPI formula - Female: 1) Serum creatinine (Scr) less than or equal to (<=)0.7 mg/dL: 144*(Scr/0.7)^-0.329*0.993age; 2) Scr greater than (>)0.7 mg/dL: 144*(Scr/0.7)^-1.209*0.993age. Male: 1) Scr <=0.9 mg/dL: 141*(Scr/0.9)^-0.411*0.993age; 2) Scr >0.9 mg/dL: 141*(Scr/0.9)^-1.209*0.993age.
Time Frame: Baseline, Weeks 24 and 48
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: mL/min/1.73 m^2
Arm/Group | D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) | Control (Baseline to Switch)
Number analyzed (Participants) | 761 | 378
mL/min/1.73 m^2
  Change at Week 24: number analyzed (Participants) | 735 | 362
  Change at Week 24 | -1.67 (0.359) | -0.75 (0.510)
  Change at Week 48: number analyzed (Participants) | 725 | 350
  Change at Week 48 | -1.97 (0.369) | -0.88 (0.531)
Statistical Analysis 1: Comparison: D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) vs Control (Baseline to Switch); Change at Week 24; Test type: Other; p = 0.143, ANCOVA; LS Mean Difference = -0.92, 95% CI 2-sided [-2.14 to 0.31], Standard Error of Mean 0.624
Statistical Analysis 2: Comparison: D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) vs Control (Baseline to Switch); Change at Week 48; Test type: Other; p = 0.092, ANCOVA; LS Mean Difference = -1.09, 95% CI 2-sided [-2.36 to 0.18], Standard Error of Mean 0.646

9. Secondary Outcome: Change From Baseline in Estimated Glomerular Filtration Rate Based on Serum Cystatin C (eGFRcyst, by Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI]) at Weeks 24 and 48
Description: Change from baseline in eGFRcyst (by CKD-EPI) was assessed at Weeks 24 and 48. eGFRcyst according to the CKD-EPI formula - 1) Serum Cystatin C (Scyst) <=0.8 mg/L: 133*(Scyst/0.8)^-0.499*0.996age (*0.932 if female); 2) Scyst >0.8 mg/L: 133*(Scyst/0.8)^-1.328*0.996age (*0.932 if female).
Time Frame: Baseline, Weeks 24 and 48
Population: ITT analysis set included all the participants who were randomized and received at least 1 dose of study treatment. Here, 'n' specifies those participants who were analyzed for this endpoint at given time point.
Measure: Least Squares Mean (Standard Error); unit: mL/min/1.73 m^2
Arm/Group | D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) | Control (Baseline to Switch)
Number analyzed (Participants) | 763 | 378
mL/min/1.73 m^2
  eGFRcyst: Change at Week 24: number analyzed (Participants) | 734 | 360
  eGFRcyst: Change at Week 24 | 0.21 (0.338) | -0.93 (0.483)
  eGFRcyst: Change at Week 48: number analyzed (Participants) | 724 | 351
  eGFRcyst: Change at Week 48 | -0.42 (0.360) | -1.76 (0.517)
Statistical Analysis 1: Comparison: D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) vs Control (Baseline to Switch); Change at Week 24; Test type: Other; p = 0.054, ANCOVA; LS Mean Difference = 1.14, 95% CI 2-sided [-0.02 to 2.29], Standard Error of Mean 0.590
Statistical Analysis 2: Comparison: D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) vs Control (Baseline to Switch); Change at Week 48; Test type: Other; p = 0.034, ANCOVA; LS Mean Difference = 1.34, 95% CI 2-sided [0.10 to 2.57], Standard Error of Mean 0.630

10. Secondary Outcome: Change From Baseline in Urine Albumin to Creatinine Ratio (UACR) and Urine Protein to Creatinine Ratio (UPCR) at Weeks 24 and 48
Description: Change from baseline in UACR and UPCR was assessed at Weeks 24 and 48. Lower levels of albumin or protein in the urine indicates better proximal tubular function.
Time Frame: Baseline, Weeks 24 and 48
Population: as for outcome 7
Measure: Median (Full Range); unit: milligram per gram (mg/g)
Arm/Group | D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) | Control (Baseline to Switch)
Number analyzed (Participants) | 761 | 378
milligram per gram (mg/g)
  UACR: Baseline | 6.20 [1.4 to 632.1] | 7.14 [1.1 to 268.0]
  UACR: Change at Week 24: number analyzed (Participants) | 735 | 362
  UACR: Change at Week 24 | -0.78 [-185.4 to 422.2] | 0.44 [-238.5 to 145.0]
  UACR: Change at Week 48: number analyzed (Participants) | 723 | 351
  UACR: Change at Week 48 | -0.76 [-195.8 to 344.3] | 0.40 [-121.7 to 110.9]
  UPCR: Baseline: number analyzed (Participants) | 758 | 375
  UPCR: Baseline | 61.56 [16.9 to 1158.1] | 62.90 [14.7 to 870.9]
  UPCR: Change at Week 24: number analyzed (Participants) | 727 | 357
  UPCR: Change at Week 24 | -14.63 [-509.6 to 734.6] | 0.07 [-359.9 to 400.8]
  UPCR: Change at Week 48: number analyzed (Participants) | 710 | 347
  UPCR: Change at Week 48 | -22.25 [-520.1 to 386.6] | -7.37 [-368.7 to 432.3]
Statistical Analysis 1: Comparison: D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) vs Control (Baseline to Switch); UACR - Change at Week 24; Test type: Other; p < 0.001, Van Elteren Test
Statistical Analysis 2: Comparison: D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) vs Control (Baseline to Switch); UACR - Change at Week 48; Test type: Other; p < 0.001, Van Elteren Test
Statistical Analysis 3: Comparison: D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) vs Control (Baseline to Switch); UPCR - Change at Week 24; Test type: Other; p < 0.001, Van Elteren Test
Statistical Analysis 4: Comparison: D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) vs Control (Baseline to Switch); UPCR - Change at Week 48; Test type: Other; p < 0.001, Van Elteren Test

11. Secondary Outcome: Change From Baseline in Urine Retinol Binding Protein to Creatinine Ratio (URBPCR) and Urine Beta-2 Microglobulin to Creatinine Ratio (UB2MGCR) at Weeks 24 and 48
Description: Change from baseline in URBPCR and UB2MGCR was assessed at Weeks 24 and 48. Retinol binding protein is a marker of proximal tubular function.
Time Frame: Baseline, Weeks 24 and 48
Population: as for outcome 7
Measure: Median (Full Range); unit: microgram per gram (mcg/g)
Arm/Group | D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) | Control (Baseline to Switch)
Number analyzed (Participants) | 748 | 371
microgram per gram (mcg/g)
  URBPCR: Baseline | 126.19 [20.3 to 116216.2] | 137.16 [12.9 to 73958.4]
  URBPCR: Change at Week 24: number analyzed (Participants) | 721 | 356
  URBPCR: Change at Week 24 | -30.27 [-69873.2 to 2004.4] | 7.76 [-6040.1 to 60740.4]
  URBPCR: Change at Week 48: number analyzed (Participants) | 710 | 344
  URBPCR: Change at Week 48 | -27.09 [-67540.0 to 1764.3] | 19.66 [-5778.3 to 65203.3]
  UB2MGCR: Baseline: number analyzed (Participants) | 736 | 366
  UB2MGCR: Baseline | 156.85 [3.8 to 91216.2] | 172.25 [9.8 to 92740.1]
  UB2MGCR: Change at Week 24: number analyzed (Participants) | 702 | 348
  UB2MGCR: Change at Week 24 | -72.64 [-72264.6 to 13536.2] | 12.08 [-20084.8 to 58357.6]
  UB2MGCR: Change at Week 48: number analyzed (Participants) | 693 | 338
  UB2MGCR: Change at Week 48 | -67.02 [-72323.4 to 21190.2] | 20.24 [-22173.5 to 135576.9]
Statistical Analysis 1: Comparison: D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) vs Control (Baseline to Switch); URBPCR: Change at Week 24; Test type: Other; p < 0.001, Van Elteren Test
Statistical Analysis 2: Comparison: D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) vs Control (Baseline to Switch); URBPCR: Change at Week 48; Test type: Other; p < 0.001, Van Elteren Test
Statistical Analysis 3: Comparison: D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) vs Control (Baseline to Switch); UB2MGCR: Change at Week 24; Test type: Other; p < 0.001, Van Elteren Test
Statistical Analysis 4: Comparison: D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) vs Control (Baseline to Switch); UB2MGCR: Change at Week 48; Test type: Other; p < 0.001, Van Elteren Test

12. Secondary Outcome: Percent Change From Baseline in Urine Fractional Excretion of Phosphate (FEPO4) at Weeks 24 and 48
Description: Percent change from baseline in urine FEPO4 was assessed at Weeks 24 and 48.
Time Frame: Baseline, Weeks 24 and 48
Population: ITT analysis set included all the participants who were randomized and received at least 1 dose of study treatment. Here 'n' specifies those participants who were analyzed for this endpoint at given time point.
Measure: Median (Full Range); unit: Percent change
Arm/Group | D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) | Control (Baseline to Switch)
Number analyzed (Participants) | 763 | 378
Percent change
  Percent change at Week 24: number analyzed (Participants) | 729 | 358
  Percent change at Week 24 | 3.58 [-89.4 to 1940.4] | 8.55 [-78.5 to 281.8]
  Percent change at Week 48: number analyzed (Participants) | 719 | 346
  Percent change at Week 48 | 8.42 [-97.9 to 1430.3] | 8.57 [-76.3 to 452.7]
Statistical Analysis 1: Comparison: D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) vs Control (Baseline to Switch); FEPO4 - Change at Week 24; Test type: Other; p = 0.288, Van Elteren Test
Statistical Analysis 2: Comparison: D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) vs Control (Baseline to Switch); FEPO4 - Change at Week 48; Test type: Other; p = 0.148, Van Elteren Test

13. Secondary Outcome: Percentage of Participants With Virologic Response Based on HIV-1 RNA Less Than (<)20, <50, and <200 Copies/mL Threshold at Week 48 as Defined by the Food and Drug Administration (FDA) Snapshot Approach
Description: Percentage of participants with virologic response based on HIV-1 RNA <20, <50, and <200 copies/mL threshold were analyzed at Week 48 using FDA snapshot approach. FDA Snapshot approach analysis was based on the last observed viral load data: virologic response was defined as HIV-1 RNA <20/50/200 copies/mL (observed case).
Time Frame: Week 48
Population: ITT analysis set included all the participants who were randomized and received at least 1 dose of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) | Control (Baseline to Switch)
Number analyzed (Participants) | 763 | 378
Percentage of Participants
  <20 copies/mL | 89.8 [87.4 to 91.8] | 88.4 [84.7 to 91.4]
  <50 copies/mL | 94.9 [93.1 to 96.3] | 93.7 [90.7 to 95.9]
  <200 copies/mL | 95.0 [93.2 to 96.5] | 94.2 [91.3 to 96.3]

14. Secondary Outcome: Percentage of Participants With Virologic Response Based on HIV-1 RNA <20, <50, and <200 Copies/mL Threshold at Week 48 as Defined by the Time to Loss of Virologic Response (TLOVR) Algorithm
Description: Percentage of participants with virologic response based on HIV-1 RNA <20, <50, and <200 copies/mL threshold were analyzed at Week 48 using TLOVR algorithm approach. TLOVR was defined as sustained HIV-1 RNA <20/50/200 copies/mL.
Time Frame: Week 48
Population: ITT analysis set included all the participants who were randomized and received at least 1 dose of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) | Control (Baseline to Switch)
Number analyzed (Participants) | 763 | 378
Percentage of Participants
  <20 copies/mL | 86.0 [83.3 to 88.4] | 83.6 [79.5 to 87.2]
  <50 copies/mL | 93.7 [91.7 to 95.3] | 92.9 [89.8 to 95.2]
  <200 copies/mL | 95.4 [93.7 to 96.8] | 94.7 [91.9 to 96.7]

15. Secondary Outcome: Change From Baseline in Cluster of Differentiation 4 Plus (CD4+) Cell Count at Weeks 24 and 48
Description: Change from baseline in CD4+ cell count was assessed at Weeks 24 and 48.
Time Frame: Baseline, Weeks 24 and 48
Population: as for outcome 12
Measure: Mean (Standard Error); unit: Cells per cubic millimeter (cells/mm^3)
Arm/Group | D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) | Control (Baseline to Switch)
Number analyzed (Participants) | 763 | 378
Cells per cubic millimeter (cells/mm^3)
  Baseline | 653.3 (9.12) | 641.7 (13.15)
  Change at Week 24: number analyzed (Participants) | 731 | 362
  Change at Week 24 | 14.3 (5.99) | 8.5 (7.76)
  Change at Week 48: number analyzed (Participants) | 722 | 351
  Change at Week 48 | 21.0 (5.97) | 9.1 (8.41)

16. Secondary Outcome: Percentage of Participants With Treatment Adherence of Greater Than (>)95 Percent (%) (Approach 1) Through Week 48
Description: Treatment adherence (defined as adherence of >95%) was assessed by the drug accountability cumulative through Week 48 (Approach 1).
Time Frame: Through Week 48
Population: ITT analysis set included all the participants who were randomized and received at least 1 dose of study treatment. Here, N (number of participants analyzed) indicates the number of participants evaluable for this endpoint.
Measure: Number; unit: Percentage of Participants
Arm/Group | D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) | Control (Baseline to Switch)
Number analyzed (Participants) | 215 | 102
Percentage of Participants | 91.6 | 85.3

17. Secondary Outcome: Percentage of Participants With Treatment Adherence of >95% (Approach 2) Through Week 48
Description: Treatment adherence (defined as adherence of >95%) was assessed by the drug accountability cumulative treatment adherence up to time point where not more than one bottle was missing, or if available, through Week 48, whichever came sooner (Approach 2).
Time Frame: Through Week 48
Population: ITT analysis set included all the participants who were randomized and received at least 1 dose of study treatment. Here, 'N' (number of participants analyzed) indicates the number of participants evaluable for this endpoint.
Measure: Number; unit: percentage of participants
Arm/Group | D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) | Control (Baseline to Switch)
Number analyzed (Participants) | 631 | 268
percentage of participants | 82.7 | 77.2

18. Secondary Outcome: Number of Participants With Resistance to Study Drug
Description: HIV-1 genotypes were analyzed from samples of participants with confirmed virologic rebound (virologic rebound was defined as: confirmed HIV-1 RNA >=50 copies/mL up to, and including the upper bound of the Week 48 window) and with HIV-1 RNA value >=400 copies/mL or who discontinued with last HIV-1 RNA >=400 copies/mL. Number of participants who developed resistance to any of the study drug was determined.
Time Frame: Up to Week 48
Population: The ITT population with confirmed virologic rebound and with HIV-1 RNA value >=400 copies/mL was analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) | Control (Baseline to Switch)
Number analyzed (Participants) | 19 | 8
Participants | 1 | 3

19. Secondary Outcome: Predose (Trough) Plasma Concentration (C0h) of Darunavir
Description: Predose (trough) plasma concentration (C0h) of darunavir was determined. Pharmacokinetic (PK) data was only analyzed for participants in the D/C/F/TAF group as per planned analysis.
Time Frame: Predose at Weeks 2, 4, 8, 12, 24, 36, and 48
Population: The PK analysis set included all participants randomized to D/C/F/TAF group and received at least 1 dose of study drug in study, and for whom plasma concentration data of any analytes of interest were available. Here 'n' specifies participants who were analyzed for this endpoint at given time point.
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter (ng/mL)
Arm/Group | D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE])
Number analyzed (Participants) | 750
Nanogram per milliliter (ng/mL)
  Week 2: number analyzed (Participants) | 130
  Week 2 | 1775.29 (1698.84)
  Week 4: number analyzed (Participants) | 110
  Week 4 | 1732.00 (1389.44)
  Week 8: number analyzed (Participants) | 104
  Week 8 | 1910.30 (1501.94)
  Week 12: number analyzed (Participants) | 114
  Week 12 | 1643.38 (1328.41)
  Week 24: number analyzed (Participants) | 112
  Week 24 | 2022.99 (1965.64)
  Week 36: number analyzed (Participants) | 100
  Week 36 | 1806.37 (1669.43)
  Week 48: number analyzed (Participants) | 126
  Week 48 | 1899.79 (1833.09)

20. Secondary Outcome: Percent Change From Baseline in Serum Procollagen 1 N-Terminal Propeptide (P1NP) and Serum Collagen Type 1 Beta Carboxy Telopeptide (CTX) Levels at Weeks 24 and 48
Description: Percent change from baseline in bone biomarkers: P1NP and CTX was assessed at Weeks 24 and 48.
Time Frame: Baseline, Weeks 24 and 48
Population: The bone investigation substudy (BIS) analysis set included all participants who were randomized and received at least 1 dose of study drug in the study, and had at least one postbaseline value for biomarker data. Here 'n' specifies participants who were analyzed for this endpoint at given time point.
Measure: Mean (Standard Error); unit: Percent Change
Arm/Group | D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) | Control (Baseline to Switch)
Number analyzed (Participants) | 209 | 108
Percent Change
  P1NP: Percent change at Week 24: number analyzed (Participants) | 195 | 99
  P1NP: Percent change at Week 24 | -22.971 (1.8818) | -0.027 (2.7325)
  P1NP: Percent change at Week 48: number analyzed (Participants) | 191 | 98
  P1NP: Percent change at Week 48 | -26.752 (1.8960) | -3.751 (2.6988)
  CTX: Percent change at Week 24: number analyzed (Participants) | 190 | 97
  CTX: Percent change at Week 24 | -16.772 (2.2575) | 16.312 (3.8855)
  CTX: Percent change at Week 48: number analyzed (Participants) | 185 | 98
  CTX: Percent change at Week 48 | -10.517 (3.2325) | 5.433 (4.1118)

21. Secondary Outcome: Percent Change From Baseline in Parathyroid Hormone (PTH) at Weeks 24 and 48
Description: Percent change from baseline in bone biomarker: PTH was assessed at Weeks 24 and 48.
Time Frame: Baseline, Weeks 24 and 48
Population: as for outcome 20
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) | Control (Baseline to Switch)
Number analyzed (Participants) | 209 | 108
Percent change
  Percent change at Week 24: number analyzed (Participants) | 199 | 102
  Percent change at Week 24 | -3.092 (2.5941) | 12.034 (4.1777)
  Percent change at Week 48: number analyzed (Participants) | 193 | 103
  Percent change at Week 48 | -4.510 (2.5375) | 9.436 (4.4784)

22. Secondary Outcome: Percent Change From Baseline in 25-hydroxy Vitamin D at Weeks 24 and 48
Description: Percent change from baseline in bone biomarker: 25-hydroxy vitamin D was assessed at Weeks 24 and 48.
Time Frame: Baseline, Weeks 24 and 48
Population: as for outcome 20
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) | Control (Baseline to Switch)
Number analyzed (Participants) | 209 | 108
Percent change
  Percent change at Week 24: number analyzed (Participants) | 146 | 72
  Percent change at Week 24 | -3.0 (5.06) | 4.2 (6.13)
  Percent change at Week 48: number analyzed (Participants) | 142 | 72
  Percent change at Week 48 | 25.2 (5.51) | 24.9 (7.46)

23. Secondary Outcome: Percent Change From Baseline in Spine and Hip Bone Mineral Density (BMD) at Weeks 24 and 48
Description: Percent change from baseline in spine and hip BMD was assessed at Weeks 24 and 48.
Time Frame: Baseline, Weeks 24 and 48
Population: The bone investigation substudy (BIS) analysis set included all participants who were randomized and received at least 1 dose of study drug in the study, and had at least one postbaseline value for bone mineral density (BMD) data. Here 'n' specifies participants who were analyzed for this endpoint at given time point.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) | Control (Baseline to Switch)
Number analyzed (Participants) | 209 | 108
Percent change
  Spine BMD: Percent change at Week 24: number analyzed (Participants) | 192 | 97
  Spine BMD: Percent change at Week 24 | 1.55 (0.276) | 0.18 (0.342)
  Spine BMD: Percent change at Week 48: number analyzed (Participants) | 192 | 101
  Spine BMD: Percent change at Week 48 | 2.06 (0.324) | 0.01 (0.391)
  Hip BMD: Percent change at Week 24: number analyzed (Participants) | 184 | 93
  Hip BMD: Percent change at Week 24 | 0.91 (0.230) | 0.00 (0.279)
  Hip BMD: Percent change at Week 48: number analyzed (Participants) | 188 | 97
  Hip BMD: Percent change at Week 48 | 1.62 (0.244) | -0.08 (0.288)
Statistical Analysis 1: Comparison: D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) vs Control (Baseline to Switch); Spine BMD: Percent change at Week 24; Test type: Other; p < 0.001, ANCOVA; LS Mean Difference = 1.37, 95% CI 2-sided [0.697 to 2.037], Standard Error of Mean 0.340
Statistical Analysis 2: Comparison: D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) vs Control (Baseline to Switch); Spine BMD: Percent change at Week 48; Test type: Other; p < 0.001, ANCOVA; LS Mean Difference = 2.05, 95% CI 2-sided [1.277 to 2.814], Standard Error of Mean 0.390
Statistical Analysis 3: Comparison: D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) vs Control (Baseline to Switch); Hip BMD: Percent change at Week 24; Test type: Other; p = 0.001, ANCOVA; LS Mean Difference = 0.90, 95% CI 2-sided [0.366 to 1.436], Standard Error of Mean 0.272
Statistical Analysis 4: Comparison: D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) vs Control (Baseline to Switch); Hip BMD: Percent change at Week 48; Test type: Other; p < 0.001, ANCOVA; LS Mean Difference = 1.70, 95% CI 2-sided [1.144 to 2.248], Standard Error of Mean 0.280

24. Secondary Outcome: Change From Baseline in Bone Mineral Density (BMD) T-Score at Weeks 24 and 48
Description: Change from baseline in spine, hip, and femoral neck BMD T-Score was assessed at Week 24 and 48. T-score values >= -1.0 were considered normal, T-score values < -1.0 to -2.5 indicate osteopenia and T-score values < -2.5 indicate osteoporosis.
Time Frame: Baseline, Weeks 24 and 48
Population: The bone investigation substudy (BIS) analysis set included all participants who were randomized and received at least 1 dose of study drug in the study, and had at least one postbaseline value for BMD data. Here 'n' specifies those participants who were analyzed for this endpoint at given time point.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) | Control (Baseline to Switch)
Number analyzed (Participants) | 209 | 108
Units on a scale
  Spine BMD T-score: Baseline: number analyzed (Participants) | 206 | 107
  Spine BMD T-score: Baseline | -0.713 (0.0850) | -0.467 (0.1260)
  Spine BMD T-score: Change at Week 24: number analyzed (Participants) | 192 | 97
  Spine BMD T-score: Change at Week 24 | 0.102 (0.0172) | -0.033 (0.0253)
  Spine BMD T-score: Change at Week 48: number analyzed (Participants) | 192 | 101
  Spine BMD T-score: Change at Week 48 | 0.132 (0.0217) | -0.063 (0.0264)
  Hip BMD T-score: Baseline: number analyzed (Participants) | 204 | 104
  Hip BMD T-score: Baseline | -0.575 (0.0643) | -0.484 (0.0839)
  Hip BMD T-score: Change at Week 24: number analyzed (Participants) | 184 | 93
  Hip BMD T-score: Change at Week 24 | 0.037 (0.0108) | -0.024 (0.0144)
  Hip BMD T-score: Change at Week 48: number analyzed (Participants) | 188 | 97
  Hip BMD T-score: Change at Week 48 | 0.095 (0.0122) | -0.016 (0.0139)
  Femoral Neck BMD T-score: Baseline: number analyzed (Participants) | 204 | 104
  Femoral Neck BMD T-score: Baseline | -0.782 (0.0625) | -0.699 (0.0899)
  Femoral Neck BMD T-score: Change at Week 24: number analyzed (Participants) | 184 | 93
  Femoral Neck BMD T-score: Change at Week 24 | 0.019 (0.0128) | -0.044 (0.0183)
  Femoral Neck BMD T-score: Change at Week 48: number analyzed (Participants) | 188 | 97
  Femoral Neck BMD T-score: Change at Week 48 | 0.039 (0.0146) | -0.039 (0.0214)

25. Secondary Outcome: Percentage of Participants With Virologic Rebound (HIV-1 RNA >=20 Copies/mL) Cumulative Through Week 96
Description: Virologic rebound was defined as: confirmed plasma HIV-1 RNA level >=20 copies/mL up to and including Week 96, last available on-treatment (single) HIV-1 RNA >=20 copies/mL at premature discontinuation (irrespective of reason), and last available on-treatment HIV-1 RNA >=20 copies/mL at the study cutoff of Week 96 (that is, any last viral load [re]test having occurred no later than 6 weeks after Week 96). Percentage of participants with virologic rebound were reported.
Time Frame: Through Week 96 (D/C/F/TAF arm) and from Week 52 to Week 96 (Switch to D/C/F/TAF arm)
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) | Switch to D/C/F/TAF
Number analyzed (Participants) | 763 | 352
percentage of participants | 13.8 [11.4 to 16.4] | 8.8 [6.1 to 12.3]

26. Secondary Outcome: Percentage of Participants With Virologic Rebound (HIV-1 RNA >=50 Copies/mL) Cumulative Through Week 96
Description: Virologic rebound was defined as: confirmed plasma HIV-1 RNA level >=50 copies/mL up to and including Week 96, last available on-treatment (single) HIV-1 RNA >=50 copies/mL at premature discontinuation (irrespective of reason), and last available on-treatment HIV-1 RNA >=50copies/mL at the study cutoff of Week 96 (that is, any last viral load [re]test having occurred no later than 6 weeks after Week 96). Percentage of participants with virologic rebound were reported.
Time Frame: Through Week 96 (D/C/F/TAF arm) and from Week 52 to Week 96 (Switch to D/C/F/TAF arm)
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) | Switch to D/C/F/TAF
Number analyzed (Participants) | 763 | 352
percentage of participants | 3.1 [2.0 to 4.6] | 2.3 [1.0 to 4.4]

27. Secondary Outcome: Percentage of Participants With Virologic Rebound (HIV-1 RNA >=200 Copies/mL) Cumulative Through Week 96
Description: Virologic rebound was defined as: confirmed plasma HIV-1 RNA level >=200 copies/mL up to and including Week 96, last available on-treatment (single) HIV-1 RNA >=200 copies/mL at premature discontinuation (irrespective of reason), and last available on-treatment HIV-1 RNA >=200 copies/mL at the study cutoff of Week 96 (that is, any last viral load [re]test having occurred no later than 6 weeks after Week 96). Percentage of participants with virologic rebound were reported.
Time Frame: Through Week 96 (D/C/F/TAF arm) and from Week 52 to Week 96 (Switch to D/C/F/TAF arm)
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) | Switch to D/C/F/TAF
Number analyzed (Participants) | 763 | 352
percentage of participants | 0.5 [0.1 to 1.3] | 0.6 [0.1 to 2.0]

28. Secondary Outcome: Percentage of Participants With Non-Virologic Rebound at Week 96 by Kaplan-Meier Estimates
Description: Here Kaplan-Meier estimates percentage of participants with non-virologic rebound at Week 96.
Time Frame: Baseline to Week 96 (D/C/F/TAF arm) and from Week 52 to Week 96 (Switch to D/C/F/TAF arm)
Population: ITT analysis set included all the participants who were randomized and received at least 1 dose of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) | Switch to D/C/F/TAF
Number analyzed (Participants) | 763 | 352
percentage of participants | 96.7 [95.1 to 97.8] | 97.8 [95.4 to 98.9]

29. Secondary Outcome: Percentage of Participants With Virologic Response Based on HIV-1 RNA <20, <50, and <200 Copies/mL Threshold at Week 96 as Defined by the FDA Snapshot Approach
Description: Percentage of participants with virologic response based on HIV-1 RNA <20, <50, and <200 copies/mL threshold were analyzed at Week 96 using FDA snapshot approach. FDA Snapshot approach analysis was based on the last observed viral load data: virologic response was defined as having last available HIV-1 RNA <20/50/200 copies/mL (observed case).
Time Frame: Week 96 (Comprising up to Week 96 for D/C/F/TAF and 44 weeks of D/C/F/TAF exposure [that is, from the switch to D/C/F/TAF at Week 52 up to Week 96])
Population: ITT analysis set included all the participants who were randomized and received at least 1 dose of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) | Switch to D/C/F/TAF
Number analyzed (Participants) | 763 | 352
percentage of participants
  <20 copies/mL | 85.3 [82.6 to 87.8] | 89.8 [86.1 to 92.7]
  <50 copies/mL | 90.7 [88.4 to 92.7] | 93.8 [90.7 to 96]
  <200 copies/mL | 91.2 [89.0 to 93.1] | 95.5 [92.7 to 97.4]

30. Secondary Outcome: Percentage of Participants With Virologic Response Based on HIV-1 RNA <20, <50, and <200 Copies/mL Threshold at Week 96 as Defined by the TLOVR Algorithm
Description: Percentage of participants with virologic response based on HIV-1 RNA <20, <50, and <200 copies/mL threshold were analyzed at Week 96 using TLOVR algorithm approach. TLOVR was defined as sustained HIV-1 RNA <20/50/200 copies/mL.
Time Frame: as for outcome 29
Population: ITT analysis set included all the participants who were randomized and received at least 1 dose of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) | Switch to D/C/F/TAF
Number analyzed (Participants) | 763 | 352
percentage of participants
  <20 copies/mL | 79.6 [76.5 to 82.4] | 88.1 [84.2 to 91.3]
  <50 copies/mL | 89.6 [87.3 to 91.7] | 94.3 [91.4 to 96.5]
  <200 copies/mL | 91.7 [89.6 to 93.6] | 95.7 [93.1 to 97.6]

31. Secondary Outcome: Percentage of Participants With Virologic Failure Based on HIV-1 RNA >=20, >=50, and >=200 Copies/mL Threshold at Week 96 as Defined by the FDA Snapshot Approach
Description: Percentage of participants with virologic failure based on HIV-1 RNA >=20, >=50, and >=200 copies/mL threshold were analyzed at Week 96 using FDA snapshot approach. FDA Snapshot approach analysis was based on the last observed viral load data: virologic failure was defined by the FDA snapshot approach as having last available HIV-1 RNA >=20/50/200 copies/mL at Week 96; virologic failure - leading to discontinuation; virologic failure - discontinued due to other reason and last available HIV-1 RNA >=20/50/200 copies/mL.
Time Frame: as for outcome 29
Population: ITT analysis set included all the participants who were randomized and received at least 1 dose of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) | Switch to D/C/F/TAF
Number analyzed (Participants) | 763 | 352
percentage of participants
  >=20 copies/mL | 6.8 [5.1 to 8.8] | 6.0 [3.7 to 9.0]
  >=50 copies/mL | 1.2 [0.5 to 2.2] | 1.7 [0.6 to 3.7]
  >=200 copies/mL | 0.3 [0.0 to 0.9] | 0 [NA to NA] — NA signifies that confidence interval was not calculated as none of the participants had HIV RNA <200 copies/mL.

32. Secondary Outcome: Change From Reference in CD4+ Cell Count at Week 96
Description: Change from reference in CD4+ cell count was assessed at Week 96. The change from reference in CD4+ count at a given time point is defined as: CD4+ at a given time point minus reference CD4+. For the D/C/F/TAF group, reference is the comparative treatment phase baseline as in Week 48 analysis (reference 1). For the Switch to D/C/F/TAF (late switch) group, the last value prior to the switch was used as reference (reference 2).
Time Frame: From Reference 1 to Week 96 for D/C/F/TAF+ F/TDF Group and Reference 2 to Week 96 for Switch to D/C/F/TAF (Comprising 44 weeks of D/C/F/TAF exposure [that is, from the switch to D/C/F/TAF at Week 52])
Population: ITT analysis set included all the participants who were randomized and received at least 1 dose of study treatment. Based on non-completing=failure (NC=F) analysis with values after discontinuation imputed with the reference value. Other (intermittent) missing values are imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: cells per cubic millimeter (cells/mm^3)
Arm/Group | D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) | Switch to D/C/F/TAF
Number analyzed (Participants) | 763 | 352
cells per cubic millimeter (cells/mm^3) | 32.07 (8.0) | 13.07 (10.7)

33. Secondary Outcome: Number of Participants With Resistance to Study Drug Through Week 96
Description: HIV-1 genotypes were analyzed from samples of participants with confirmed virologic rebound in case they had HIV-1 RNA values >=400 copies/mL at failure or at later time points, including participants who discontinued with last HIV-1 RNA >=400 copies/mL. Virologic rebound was defined as: confirmed plasma HIV-1 RNA level >=20 copies/mL up to and including Week 96, last available on-treatment (single) HIV-1 RNA >=20 copies/mL at premature discontinuation (irrespective of reason), and last available on-treatment HIV-1 RNA >=20 copies/mL at the study cutoff of Week 96 (that is, any last viral load [re]test having occurred no later than 6 weeks after Week 96). Number of participants who developed resistance to any of the study drug (DRV, FTC, and TFV/TAF) were reported.
Time Frame: Through Week 96 (D/C/F/TAF arm), up to Week 48 (Control arm) and from Week 52 to Week 96 (Switch to D/C/F/TAF arm)
Population: The ITT analysis set included all the participants who were randomized and received at least one dose of study treatment in the study. Here, N (number of participants analyzed) signifies total number of participants with screening/baseline and endpoint genotype. Due to the low proportion of rebounders of which the majority had low viral load values, few samples were eligible for postbaseline genotyping.
Measure: Count of Participants; unit: Participants
Arm/Group | D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) | Control (Baseline to Switch) | Switch to D/C/F/TAF
Number analyzed (Participants) | 9 | 3 | 7
Participants
  DRV resistance-associated mutations (RAMs) | 0 | 0 | 0
  TFV RAMs | 0 | 0 | 0
  FTC RAMs | 0 | 0 | 1

34. Secondary Outcome: Percentage of Participants With Treatment Adherence of >95 (Approach 1) Through Week 96
Description: Treatment adherence (defined as adherence of >95%) was assessed by the drug accountability cumulative through Week 96 (Approach 1).
Time Frame: Through Week 96 (D/C/F/TAF arm) and from Week 52 to Week 96 (Switch to D/C/F/TAF arm)
Population: ITT analysis set included all the participants who were randomized and received at least 1 dose of study treatment. Here, N (number of participants analyzed) indicates the number of participants evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) | Switch to D/C/F/TAF
Number analyzed (Participants) | 379 | 236
percentage of participants | 91.6 | 87.3

35. Secondary Outcome: Percentage of Participants With Treatment Adherence of >95% (Approach 2) Through Week 96
Description: Treatment adherence (defined as adherence of >95%) was assessed by the drug accountability cumulative treatment adherence up to time point where not more than one bottle was missing, or if available, through Week 96, whichever came sooner (Approach 2).
Time Frame: Through Week 96 (D/C/F/TAF arm) and from Week 52 to Week 96 (Switch to D/C/F/TAF arm)
Population: ITT analysis set included all the participants who were randomized and received at least 1 dose of study treatment. Here, 'N' (number of participants analyzed) indicates the number of participants evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) | Switch to D/C/F/TAF
Number analyzed (Participants) | 646 | 320
percentage of participants | 82.8 | 80.9

36. Secondary Outcome: Percentage of Participants Experiencing Grade 3 and Grade 4 AEs, SAEs, and Premature Discontinuation Due to AEs Through Week 96
Description: AE is any untoward medical occurrence in participant who received study drug without regard to possibility of causal relationship. Grade 3 (Severe) events were symptoms causing inability to perform usual social & functional activities. Grade 4 (Life-threatening) events were symptoms causing inability to perform basic self-care functions or medical or operative intervention indicated to prevent permanent impairment, persistent disability, or death. SAE is any AE that results in: death, persistent or significant disability/incapacity, requires inpatient hospitalization or prolongation of existing hospitalization, is life-threatening experience, is a congenital anomaly/birth defect and may jeopardize participant and/or may require medical or surgical intervention to prevent one of the outcomes listed above.
Time Frame: Through Week 96 (D/C/F/TAF arm) and from Week 52 to Week 96 (Switch to D/C/F/TAF arm)
Population: ITT analysis set included all the participants who were randomized and received at least 1 dose of study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) | Switch to D/C/F/TAF
Number analyzed (Participants) | 763 | 352
percentage of participants
  Grade 3 AEs | 10.5 | 6.3
  Grade 4 AEs | 2.4 | 1.1
  SAEs | 8.7 | 6.0
  Premature discontinuations due to AEs | 2.2 | 2.0

37. Secondary Outcome: Change From Reference in Serum Creatinine Levels at Week 96
Description: Change from reference in serum creatinine levels at Week 96 was assessed. For the D/C/F/TAF group, reference is the comparative treatment phase baseline as in Week 48 analysis (Reference 1). For the Switch to D/C/F/TAF (late switch) group, the last value prior to the switch was used as reference (reference 2).
Time Frame: From Reference 1 to Week 96 for D/C/F/TAF+ F/TDF Group and Reference 2 to Week 96 for Switch to D/C/F/TAF
Population: The ITT analysis set included all the participants who were randomized and received at least one dose of study treatment. Here, N (number of participants analyzed) signifies participants evaluated for this outcome measure.
Measure: Median (Full Range); unit: micro mole per liter
Arm/Group | D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) | Switch to D/C/F/TAF
Number analyzed (Participants) | 692 | 336
micro mole per liter | 0.0 [-35 to 44] | 0.0 [-45 to 29]

38. Secondary Outcome: Change From Reference in Estimated Glomerular Filtration Rate Based on Serum Creatinine (eGFRcr, by Cockcroft-Gault Formula [eGFRcg]) at Week 96
Description: Change from reference in eGFRcr (by Cockcroft-Gault formula) was assessed at Week 96. eGFRcr according to the Cockcroft Gault formula- Male: (140 - age in years)*(weight in kilogram [kg])/72*(serum creatinine in milligram per deciliter [mg/dL])=eGFRcr (milliliter per minute [mL/min]); Female: (140 - age in years)*(weight in kg)/72*(serum creatinine in mg/dL)*0.85=eGFRcr (mL/min). For the D/C/F/TAF group, reference is the comparative treatment phase baseline as in Week 48 analysis (Reference 1). For the Switch to D/C/F/TAF (late switch) group, the last value prior to the switch was used as reference (reference 2).
Time Frame: From Reference 1 to Week 96 for D/C/F/TAF+ F/TDF Group and Reference 2 to Week 96 for Switch to D/C/F/TAF
Population: The ITT analysis set included all the participants who were randomized and received at least one dose of study treatment in the study. Here, N (number of participants analyzed) signifies participants evaluated for this outcome measure.
Measure: Median (Full Range); unit: milliliter per minute (mL/min)
Arm/Group | D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) | Switch to D/C/F/TAF
Number analyzed (Participants) | 692 | 336
milliliter per minute (mL/min) | -0.9 [-65 to 58] | 0.0 [-44 to 157]

39. Secondary Outcome: Change From Reference in Estimated Glomerular Filtration Rate Based on Serum Creatinine (by CKD-EPI) at Week 96
Description: Change from reference in eGFRcr (by CKD-EPI) was assessed at Week 96. eGFRcr per CKD-EPI formula - Female: 1) Serum creatinine (Scr) less than or equal to (<=)0.7 mg/dL: 144*(Scr/0.7)^-0.329*0.993^age; 2) Scr greater than (>)0.7 mg/dL: 144*(Scr/0.7)^-1.209*0.993^age. Male: 1) Scr <=0.9 mg/dL: 141*(Scr/0.9)^-0.411*0.993^age; 2) Scr >0.9 mg/dL: 141*(Scr/0.9)^-1.209*0.993^age. . For the D/C/F/TAF group, reference is the comparative treatment phase baseline as in Week 48 analysis (Reference 1). For the Switch to D/C/F/TAF (late switch) group, the last value prior to the switch was used as reference (reference 2).
Time Frame: From Reference 1 to Week 96 for D/C/F/TAF+ F/TDF Group and Reference 2 to Week 96 for Switch to D/C/F/TAF
Population: The ITT analysis set included all the participants who were randomized and participants at least one dose of study treatment. Here, N (number of participants analyzed) signifies participants evaluated for this outcome measure.
Measure: Median (Full Range); unit: mL/min/1.73 m^2
Arm/Group | D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) | Switch to D/C/F/TAF
Number analyzed (Participants) | 692 | 336
mL/min/1.73 m^2 | -1.3 [-37 to 35] | -0.7 [-31 to 49]

40. Secondary Outcome: Change From Reference in Estimated Glomerular Filtration Rate Based on Serum Cystatin C (by CKD-EPI) at Week 96
Description: Change from reference in eGFRcyst (by CKD-EPI) was assessed at Week 96. eGFRcyst according to the CKD-EPI formula - 1) Serum Cystatin C (Scyst) <=0.8 mg/L: 133*(Scyst/0.8)^-0.499*0.996^age (*0.932 if female); 2) Scyst >0.8 mg/L: 133*(Scyst/0.8)^-1.328*0.996^age (*0.932 if female). For the D/C/F/TAF group, reference is the comparative treatment phase baseline as in Week 48 analysis (Reference 1). For the Switch to D/C/F/TAF (late switch) group, the last value prior to the switch was used as reference (reference 2).
Time Frame: From Reference 1 to Week 96 for D/C/F/TAF+ F/TDF Group and Reference 2 to Week 96 for Switch to D/C/F/TAF
Population: as for outcome 39
Measure: Median (Full Range); unit: mL/min/1.73 m^2
Arm/Group | D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) | Switch to D/C/F/TAF
Number analyzed (Participants) | 686 | 332
mL/min/1.73 m^2 | -0.9 [-42 to 30] | 1.0 [-30 to 105]

41. Secondary Outcome: Change From Reference in UACR at Week 96
Description: Change from reference in UACR was assessed at Week 96. For the D/C/F/TAF group, reference is the comparative treatment phase baseline as in Week 48 analysis (Reference 1). For the Switch to D/C/F/TAF (late switch) group, the last value prior to the switch was used as reference (reference 2).
Time Frame: From Reference 1 to Week 96 for D/C/F/TAF+ F/TDF Group and Reference 2 to Week 96 for Switch to D/C/F/TAF
Population: as for outcome 37
Measure: Median (Full Range); unit: milligram per gram (mg/g)
Arm/Group | D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) | Switch to D/C/F/TAF
Number analyzed (Participants) | 694 | 334
milligram per gram (mg/g) | -0.63 [-209.3 to 2019.7] | -0.93 [-234.6 to 13230.9]

42. Secondary Outcome: Change From Reference in URBPCR at Week 96
Description: Change from reference in URBPCR was assessed at Week 96. For the D/C/F/TAF group, reference is the comparative treatment phase baseline as in Week 48 analysis (Reference 1). For the Switch to D/C/F/TAF (late switch) group, the last value prior to the switch was used as reference (reference 2).
Time Frame: From Reference 1 to Week 96 for D/C/F/TAF+ F/TDF Group and Reference 2 to Week 96 for Switch to D/C/F/TAF
Population: as for outcome 37
Measure: Median (Full Range); unit: microgram per gram (mcg/g)
Arm/Group | D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) | Switch to D/C/F/TAF
Number analyzed (Participants) | 675 | 331
microgram per gram (mcg/g) | -25.08 [-61980.5 to 1393.0] | -39.07 [-82240.7 to 869.9]

43. Secondary Outcome: Change From Reference in UPCR at Week 96
Description: Change from reference in UPCR was assessed at Week 96. For the D/C/F/TAF group, reference is the comparative treatment phase baseline as in Week 48 analysis (Reference 1). For the Switch to D/C/F/TAF (late switch) group, the last value prior to the switch was used as reference (reference 2).
Time Frame: From Reference 1 to Week 96 for D/C/F/TAF+ F/TDF Group and Reference 2 to Week 96 for Switch to D/C/F/TAF
Population: as for outcome 37
Measure: Median (Full Range); unit: milligram per gram (mg/g)
Arm/Group | D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) | Switch to D/C/F/TAF
Number analyzed (Participants) | 675 | 331
milligram per gram (mg/g) | -22.23 [-533.3 to 2314.7] | -12.81 [-722.1 to 453.1]

44. Secondary Outcome: Change From Reference in UB2MGCR at Week 96
Description: Change from reference in UB2MGCR was assessed at Week 96. For the D/C/F/TAF group, reference is the comparative treatment phase baseline as in Week 48 analysis (Reference 1). For the Switch to D/C/F/TAF (late switch) group, the last value prior to the switch was used as reference (reference 2).
Time Frame: From Reference 1 to Week 96 for D/C/F/TAF+ F/TDF Group and Reference 2 to Week 96 for Switch to D/C/F/TAF
Population: as for outcome 37
Measure: Median (Full Range); unit: microgram per gram (mcg/g)
Arm/Group | D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) | Switch to D/C/F/TAF
Number analyzed (Participants) | 664 | 332
microgram per gram (mcg/g) | -68.22 [-71549.3 to 7433.1] | -110.31 [-152500.2 to 12288.4]

45. Secondary Outcome: Percent Change From Reference in FEPO4 at Week 96
Description: Percent change from reference in FEPO4 at Week 96 was reported. For the D/C/F/TAF group, reference is the comparative treatment phase baseline as in Week 48 analysis (Reference 1). For the Switch to D/C/F/TAF (late switch) group, the last value prior to the switch was used as reference (reference 2).
Time Frame: From Reference 1 to Week 96 for D/C/F/TAF+ F/TDF Group and Reference 2 to Week 96 for Switch to D/C/F/TAF
Population: as for outcome 37
Measure: Median (Full Range); unit: percent change
Arm/Group | D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) | Switch to D/C/F/TAF
Number analyzed (Participants) | 688 | 334
percent change | 4.15 [-88.0 to 524.8] | -3.19 [-77.9 to 547.8]

46. Secondary Outcome: Percent Change From Reference in Levels of Serum P1NP at Week 96
Description: Percent change from reference in serum P1NP levels at Week 96 was reported. For the D/C/F/TAF group, reference is the comparative treatment phase baseline as in Week 48 analysis (Reference 1). For the Switch to D/C/F/TAF (late switch) group, the last value prior to the switch was used as reference (reference 2).
Time Frame: From Reference 1 to Week 96 for D/C/F/TAF+ FTC/TDF Group and Reference 2 to Week 96 for Switch to D/C/F/TAF
Population: BIS analysis set included all participants who were randomized, received at least 1 dose of study drug in study and had at least one post-baseline value for either biomarker/BMD data. Here, N (number of participants analyzed) signifies participants evaluated for this outcome measure.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) | Switch to D/C/F/TAF
Number analyzed (Participants) | 183 | 96
percent change | -19.899 (2.2151) | -18.466 (3.1169)

47. Secondary Outcome: Percent Change From Reference in Levels of Serum CTX at Week 96
Description: Percent change from reference in serum CTX at Week 96 was reported. For the D/C/F/TAF group, reference is the comparative treatment phase baseline as in Week 48 analysis (Reference 1). For the Switch to D/C/F/TAF (late switch) group, the last value prior to the switch was used as reference (reference 2).
Time Frame: From Reference 1 to Week 96 for D/C/F/TAF+ FTC/TDF Group and Reference 2 to Week 96 for Switch to D/C/F/TAF
Population: as for outcome 46
Measure: Mean (Standard Error); unit: percent change
Arm/Group | D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) | Switch to D/C/F/TAF
Number analyzed (Participants) | 178 | 98
percent change | -10.192 (3.0592) | -21.755 (3.4926)

48. Secondary Outcome: Percent Change From Reference in Levels of PTH at Week 96
Description: Percent change from reference in PTH at Week 96 was reported. For the D/C/F/TAF group, reference is the comparative treatment phase baseline as in Week 48 analysis (Reference 1). For the Switch to D/C/F/TAF (late switch) group, the last value prior to the switch was used as reference (reference 2).
Time Frame: From Reference 1 to Week 96 for D/C/F/TAF+ FTC/TDF Group and Reference 2 to Week 96 for Switch to D/C/F/TAF
Population: as for outcome 46
Measure: Mean (Standard Error); unit: percent change
Arm/Group | D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) | Switch to D/C/F/TAF
Number analyzed (Participants) | 169 | 97
percent change | -17.171 (2.6774) | -20.466 (3.2559)

49. Secondary Outcome: Percent Change From Reference in Levels of 25-OH Vitamin D at Week 96
Description: Percent change from reference in 25-OH Vitamin D at Week 96 were reported. For the D/C/F/TAF group, reference is the comparative treatment phase baseline as in Week 48 analysis (Reference 1). For the Switch to D/C/F/TAF (late switch) group, the last value prior to the switch was used as reference (reference 2).
Time Frame: From Reference 1 to Week 96 for D/C/F/TAF+ FTC/TDF Group and Reference 2 to Week 96 for Switch to D/C/F/TAF
Population: as for outcome 46
Measure: Mean (Standard Error); unit: percent change
Arm/Group | D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) | Switch to D/C/F/TAF
Number analyzed (Participants) | 141 | 98
percent change | 24.6 (5.16) | -1.9 (3.33)

50. Secondary Outcome: Percent Change From Reference in Hip and Spine BMD at Week 96
Description: The BMD is the amount of mineral in gram per square centimeter of bone, which was assessed by DXA scan. Positive values are "best values" and negative values are "worst values" of change. Percent change from reference in hip and spine BMD was assessed. For the D/C/F/TAF group, reference is the comparative treatment phase baseline as in Week 48 analysis (Reference 1). For the Switch to D/C/F/TAF (late switch) group, the last value prior to the switch was used as reference (reference 2).
Time Frame: From Reference 1 to Week 96 for D/C/F/TAF+ FTC/TDF Group and Reference 2 to Week 96 for Switch to D/C/F/TAF
Population: BIS analysis set included all participants who were randomized, received at least 1 dose of study drug in study and had at least one post-baseline value for either biomarker/BMD data. Here, N (number of participants analyzed) indicates number of participants evaluable for this outcome measure; and 'n' specifies participants analyzed for specified categories.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) | Switch to D/C/F/TAF
Number analyzed (Participants) | 173 | 99
percent change
  Hip region BMD-T score: number analyzed (Participants) | 164 | 96
  Hip region BMD-T score | 0.0173 (0.00217) | 0.0108 (0.00328)
  Spine region BMD-T score | 0.0193 (0.00286) | 0.0279 (0.00381)

51. Secondary Outcome: Change From Reference in BMD T-score of Hip and Spine at Week 96
Description: BMD status was assessed using BMD T-scores; normal bone status was defined by a BMD T-score >= -1, osteopenia by a T-score >= -2.5 to <-1.0, and osteoporosis by a T-score <-2.5. For the D/C/F/TAF group, reference is the comparative treatment phase baseline as in Week 48 analysis (Reference 1). For the Switch to D/C/F/TAF (late switch) group, the last value prior to the switch was used as reference (reference 2).
Time Frame: From Reference 1 to Week 96 for D/C/F/TAF+ FTC/TDF Group and Reference 2 to Week 96 for Switch to D/C/F/TAF
Population: as for outcome 50
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) | Switch to D/C/F/TAF
Number analyzed (Participants) | 173 | 99
units on a scale
  Hip region BMD: number analyzed (Participants) | 164 | 96
  Hip region BMD | 0.122 (0.0154) | 0.077 (0.0230)
  Spine region BMD | 0.176 (0.0259) | 0.255 (0.0339)

52. Secondary Outcome: Percentage of Participants With Non-Virologic Rebound by Kaplan-Meier Estimates
Description: Virologic rebound is defined as participants who show confirmed HIV-1 RNA >=50 copies/mL, or for which the last available (single) HIV-1 RNA value on treatment was >=50 copies/mL. Here, Kaplan-Meier estimates (%) of non-virologic rebound at every 6 months interval are presented.
Time Frame: Week 96 to end of extension (at every 6 months, up to 42 months)
Population: ITT analysis set included all the participants who were randomized and received at least 1 dose of study treatment. Here, N (number of participants analyzed) indicates number of participants evaluable for this outcome measure; and 'n' specifies participants analyzed for specified timepoints.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) | Switch to D/C/F/TAF
Number analyzed (Participants) | 671 | 323
percentage of participants
  Week 96 | 100 [100 to 100] | 100 [100 to 100]
  Week 96 + 6 months: number analyzed (Participants) | 638 | 308
  Week 96 + 6 months | 99.4 [98.4 to 99.8] | 100 [100 to 100]
  Week 96 + 12 months: number analyzed (Participants) | 515 | 248
  Week 96 + 12 months | 98.0 [96.5 to 98.9] | 98.5 [96.0 to 99.4]
  Week 96 + 18 months: number analyzed (Participants) | 325 | 159
  Week 96 + 18 months | 97.6 [95.9 to 98.6] | 98.1 [95.4 to 99.2]
  Week 96 + 24 months: number analyzed (Participants) | 150 | 68
  Week 96 + 24 months | 97.1 [94.9 to 98.3] | 96.5 [92.3 to 98.4]
  Week 96 + 30 months: number analyzed (Participants) | 55 | 28
  Week 96 + 30 months | 95.3 [91.3 to 97.5] | 96.5 [92.3 to 98.4]
  Week 96 + 36 months: number analyzed (Participants) | 26 | 8
  Week 96 + 36 months | 92.4 [83 to 96.7] | 96.5 [92.3 to 98.4]
  Week 96 + 42 months: number analyzed (Participants) | 2 | 0
  Week 96 + 42 months | 92.4 [83.0 to 96.7] |

53. Secondary Outcome: Percentage of Participants With Non-Treatment Failure by Kaplan-Meier Estimates
Description: Percentage of participants with non-treatment failure by Kaplan-Meier Estimates were reported. Treatment failure was defined as having either protocol-defined virologic rebound or having discontinued for reasons other than alternate access to D/C/F/TAF (or other antiretroviral [ARV]).
Time Frame: Week 96 to end of extension (up to 42 months)
Population: The ITT analysis set included all the participants who were randomized and received at least one dose of study treatment. Here, N (number of participants analyzed) indicates number of participants evaluable for this outcome measure; and 'n' specifies participants analyzed for specified timepoints.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) | Switch to D/C/F/TAF
Number analyzed (Participants) | 680 | 326
percentage of participants
  Week 96 | 100 [100 to 100] | 100 [100 to 100]
  Week 96 + 6 months: number analyzed (Participants) | 646 | 311
  Week 96 + 6 months | 98.1 [96.7 to 98.9] | 98.5 [96.3 to 99.4]
  Week 96 + 12 months: number analyzed (Participants) | 532 | 261
  Week 96 + 12 months | 94.3 [92.2 to 95.9] | 95.4 [92.3 to 97.2]
  Week 96 + 18 months: number analyzed (Participants) | 348 | 177
  Week 96 + 18 months | 91.6 [89.0 to 93.6] | 92.2 [88.3 to 94.8]
  Week 96 + 24 months: number analyzed (Participants) | 163 | 71
  Week 96 + 24 months | 89.4 [86.1 to 91.9] | 89.7 [85.0 to 93.0]
  Week 96 + 30 months: number analyzed (Participants) | 62 | 32
  Week 96 + 30 months | 87.0 [82.7 to 90.4] | 88.1 [82.0 to 92.2]
  Week 96 + 36 months: number analyzed (Participants) | 32 | 12
  Week 96 + 36 months | 84.9 [78.2 to 89.6] | 82.6 [67.4 to 91.1]
  Week 96 + 42 months: number analyzed (Participants) | 2 | 0
  Week 96 + 42 months | 81.7 [71.9 to 88.4] |

54. Secondary Outcome: Percentage of Participants With HIV RNA <50, <20, <200 Copies/mL Post Week 96 to End of Extension
Description: Percentage of participants with HIV RNA <50, <20, <200 copies/mL post Week 96 to end of extension were reported.
Time Frame: Week 96 to end of extension (up to 42 months)
Population: The ITT analysis set included all the participants who were randomized and received at least one dose of study treatment in the study. Here, N (number of participants analyzed) indicates number of participants evaluable for this outcome measure and 'n' specifies participants analyzed for specified timepoints.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) | Switch to D/C/F/TAF
Number analyzed (Participants) | 688 | 334
percentage of participants
  Week 96 + 6 months (<50 copies/mL) | 97.8 [96.4 to 98.8] | 97.9 [95.7 to 99.2]
  Week 96 + 12 months (<50 copies/mL): number analyzed (Participants) | 611 | 302
  Week 96 + 12 months (<50 copies/mL) | 98.4 [97.0 to 99.2] | 97.4 [94.8 to 98.8]
  Week 96 + 18 months (<50 copies/mL): number analyzed (Participants) | 461 | 225
  Week 96 + 18 months (<50 copies/mL) | 99.6 [98.4 to 99.9] | 98.7 [96.2 to 99.7]
  Week 96 + 24 months (<50 copies/mL): number analyzed (Participants) | 280 | 134
  Week 96 + 24 months (<50 copies/mL) | 99.3 [97.4 to 99.9] | 98.5 [94.7 to 99.8]
  Week 96 + 30 months (<50 copies/mL): number analyzed (Participants) | 135 | 64
  Week 96 + 30 months (<50 copies/mL) | 99.3 [95.9 to 100] | 100 [94.4 to 100]
  Week 96 + 36 months (<50 copies/mL): number analyzed (Participants) | 52 | 26
  Week 96 + 36 months (<50 copies/mL) | 98.1 [89.7 to 100] | 100 [86.8 to 100]
  Week 96 + 42 months (<50 copies/mL): number analyzed (Participants) | 16 | 7
  Week 96 + 42 months (<50 copies/mL) | 100 [79.4 to 100] | 100 [59.0 to 100]
  Week 96 + 6 months (<200 copies/mL) | 99.1 [98.1 to 99.7] | 99.7 [98.3 to 100]
  Week 96 + 12 months (<200 copies/mL): number analyzed (Participants) | 611 | 302
  Week 96 + 12 months (<200 copies/mL) | 99.3 [98.3 to 99.8] | 98.7 [96.6 to 99.6]
  Week 96 + 18 months (<200 copies/mL): number analyzed (Participants) | 461 | 225
  Week 96 + 18 months (<200 copies/mL) | 100 [99.2 to 100] | 99.1 [96.8 to 99.9]
  Week 96 + 24 months (<200 copies/mL): number analyzed (Participants) | 280 | 134
  Week 96 + 24 months (<200 copies/mL) | 99.6 [98.0 to 100] | 99.3 [95.9 to 100]
  Week 96 + 30 months (<200 copies/mL): number analyzed (Participants) | 135 | 64
  Week 96 + 30 months (<200 copies/mL) | 100 [97.3 to 100] | 100 [94.4 to 100]
  Week 96 + 36 months (<200 copies/mL): number analyzed (Participants) | 52 | 26
  Week 96 + 36 months (<200 copies/mL) | 100 [93.2 to 100] | 100 [86.8 to 100]
  Week 96 + 42 months (<200 copies/mL): number analyzed (Participants) | 16 | 7
  Week 96 + 42 months (<200 copies/mL) | 100 [79.4 to 100] | 100 [59 to 100]
  Week 96 + 6 months (<20 copies/mL) | 91.4 [89.1 to 93.4] | 93.4 [90.2 to 95.8]
  Week 96 + 12 months (<20 copies/mL): number analyzed (Participants) | 611 | 302
  Week 96 + 12 months (<20 copies/mL) | 93.9 [91.7 to 95.7] | 91.4 [87.6 to 94.3]
  Week 96 + 18 months (<20 copies/mL): number analyzed (Participants) | 461 | 225
  Week 96 + 18 months (<20 copies/mL) | 96.1 [93.9 to 97.7] | 92.9 [88.7 to 95.9]
  Week 96 + 24 months (<20 copies/mL): number analyzed (Participants) | 280 | 134
  Week 96 + 24 months (<20 copies/mL) | 96.1 [93.1 to 98.0] | 95.5 [90.5 to 98.3]
  Week 96 + 30 months (<20 copies/mL): number analyzed (Participants) | 135 | 64
  Week 96 + 30 months (<20 copies/mL) | 95.6 [90.6 to 98.4] | 92.2 [82.7 to 97.4]
  Week 96 + 36 months (<20 copies/mL): number analyzed (Participants) | 52 | 26
  Week 96 + 36 months (<20 copies/mL) | 94.2 [84.1 to 98.8] | 96.2 [80.4 to 99.9]
  Week 96 + 42 months (<20 copies/mL): number analyzed (Participants) | 16 | 7
  Week 96 + 42 months (<20 copies/mL) | 93.8 [69.8 to 99.8] | 100 [59 to 100]

55. Secondary Outcome: CD4+ Cell Count Post-Week 96 to End of Extension
Description: The immunologic change was determined by Cluster of CD4+ cell count. CD4+ cell count post-Week 96 to end of extension were assessed.
Time Frame: Week 96 to end of extension (up to 42 months)
Population: The ITT analysis set included all the participants who were randomized and received at least one dose of study treatment in the study. Here, N (number of participants analyzed) signifies participants evaluated for this outcome measure and n (number analyzed) signifies participants analyzed at specified timepoints
Measure: Mean (Standard Error); unit: cells/mm^3
Arm/Group | D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) | Switch to D/C/F/TAF
Number analyzed (Participants) | 682 | 332
cells/mm^3
  Week 96 + 6 months | 706.4 (10.51) | 681.3 (14.99)
  Week 96 + 12 months: number analyzed (Participants) | 606 | 298
  Week 96 + 12 months | 707.6 (11.93) | 676.2 (14.57)
  Week 96 + 18 months: number analyzed (Participants) | 459 | 225
  Week 96 + 18 months | 713.3 (12.16) | 686.1 (17.05)
  Week 96 + 24 months: number analyzed (Participants) | 278 | 128
  Week 96 + 24 months | 712.7 (15.98) | 686.4 (21.20)
  Week 96 + 30 months: number analyzed (Participants) | 134 | 63
  Week 96 + 30 months | 730.4 (23.24) | 685.8 (28.61)
  Week 96 + 36 months: number analyzed (Participants) | 52 | 25
  Week 96 + 36 months | 732.0 (33.10) | 733.3 (54.73)
  Week 96 + 42 months: number analyzed (Participants) | 16 | 7
  Week 96 + 42 months | 714.3 (56.26) | 705.6 (112.99)

56. Secondary Outcome: Percentage of Participants With Treatment Adherence of >95% From Week 96 to End of Extension
Description: Treatment adherence (defined as adherence of >95%) was assessed by the drug accountability and was calculated cumulative from start of treatment/switch to last study drug intake by determination of the cumulative treatment adherence in participants who returned all dispensed bottles prior to or at the last visit in the study from Week 96 to end of extension.
Time Frame: Week 96 to end of extension (up to 42 months)
Population: as for outcome 34
Measure: Number; unit: percentage of participants
Arm/Group | D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) | Switch to D/C/F/TAF
Number analyzed (Participants) | 363 | 216
percentage of participants | 89.5 | 89.4

57. Secondary Outcome: Percentage of Participants Experiencing Grade 3 and 4 AEs, Serious Adverse Events (SAEs), and Premature Discontinuation Due to AEs Post-Week 96 to End of Extension
Description: as for outcome 36
Time Frame: From Week 96 to end of extension (up to 42 months)
Population: ITT analysis set included all the participants who were randomized and received at least 1 dose of study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | D/C/F/TAF (Test) (Baseline [BL] to End of Extension [EOE]) | Switch to D/C/F/TAF
Number analyzed (Participants) | 699 | 337
percentage of participants
  Grade 3 AEs | 5.7 | 5.0
  Grade 4 AEs | 2.1 | 1.5
  SAEs | 7.3 | 7.7
  Premature discontinuations due to AEs | 1.1 | 2.1

ADVERSE EVENTS:
Time Frame: Up to 5 years and 4 months
Description: Safety was performed using intent-to-treat (ITT) analysis set included all the participants who were randomized and received at least one dose of study treatment in the study.
Groups:
- D/C/F/TAF (Test) (Baseline to End of Extension [EOE]): Participants received a single fixed dose combination (FDC) tablet containing darunavir (DRV) 800 milligram (mg)/ cobicistat (COBI) 150 mg/ emtricitabine (FTC) 200 mg/ tenofovir alafenamide (TAF) 10 mg (D/C/F/TAF tablet), orally once daily up to Week 48. After Week 48, all participants continued to receive D/C/F/TAF treatment (that is, initial switch to D/C/F/TAF group) up to Week 96. After Week 96, participants were given the opportunity to continue D/C/F/TAF treatment until the D/C/F/TAF became commercially available up to 42 months
- Switch to D/C/F/TAF Group: After Week 52, participants earlier receiving treatment with bPI+F/TDF switched to D/C/F/TAF up to Week 96. After Week 96, participants were given the opportunity to continue D/C/F/TAF treatment until the D/C/F/TAF became commercially available for up to 42 months.
Arm/Group | D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) | Control (Baseline to Switch) | Switch to D/C/F/TAF Group
All-Cause Mortality (participants affected / at risk) | 4/763 | 0/378 | 1/352
Serious Adverse Events (participants affected / at risk) | 114/763 | 18/378 | 42/352
Other Adverse Events (participants affected / at risk) | 584/763 | 222/378 | 213/352
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) (N=763) | Control (Baseline to Switch) (N=378) | Switch to D/C/F/TAF Group (N=352)
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0
Angina unstable (Cardiac disorders) | 1 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0 | 1
Myocardial infarction (Cardiac disorders) | 4 | 1 | 1
Ventricular tachycardia (Cardiac disorders) | 1 | 0 | 0
Cushing's syndrome (Endocrine disorders) | 0 | 0 | 1
Abdominal adhesions (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 1 | 0 | 0
Anal fistula (Gastrointestinal disorders) | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 1
Inflammatory bowel disease (Gastrointestinal disorders) | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Oesophageal rupture (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0
Peptic ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Rectal perforation (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Brain death (General disorders) | 1 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 0
Hernia (General disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 2 | 0 | 2
Pyrexia (General disorders) | 1 | 0 | 1
Surgical failure (General disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Hepatitis acute (Hepatobiliary disorders) | 0 | 1 | 0
Jarisch-Herxheimer reaction (Immune system disorders) | 0 | 0 | 1
Abdominal abscess (Infections and infestations) | 0 | 0 | 1
Abscess limb (Infections and infestations) | 0 | 1 | 0
Abscess oral (Infections and infestations) | 1 | 0 | 0
Anal abscess (Infections and infestations) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 2 | 0 | 3
Appendicitis perforated (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 2 | 1 | 2
Colon gangrene (Infections and infestations) | 0 | 0 | 1
Diarrhoea infectious (Infections and infestations) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 4 | 0 | 0
Epididymitis (Infections and infestations) | 0 | 1 | 0
Escherichia sepsis (Infections and infestations) | 0 | 0 | 1
Fournier's gangrene (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 4 | 0 | 0
Gastroenteritis shigella (Infections and infestations) | 1 | 0 | 0
Groin abscess (Infections and infestations) | 1 | 0 | 0
Hepatitis A (Infections and infestations) | 1 | 0 | 1
Herpes simplex meningitis (Infections and infestations) | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 1 | 0
Infectious pleural effusion (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Lymphogranuloma venereum (Infections and infestations) | 1 | 0 | 0
Malaria (Infections and infestations) | 0 | 0 | 1
Orchitis (Infections and infestations) | 0 | 0 | 1
Perineal abscess (Infections and infestations) | 0 | 1 | 1
Peritonitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 10 | 0 | 3
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0
Secondary syphilis (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 2
Septic shock (Infections and infestations) | 1 | 0 | 1
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0
Syphilis (Infections and infestations) | 0 | 1 | 0
Tooth infection (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Urosepsis (Infections and infestations) | 1 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 3 | 0 | 0
Eye injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Foreign body in gastrointestinal tract (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ligament injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 1 | 0 | 0
Musculoskeletal injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 3 | 0 | 1
Postoperative ileus (Injury, poisoning and procedural complications) | 1 | 0 | 0
Skull fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Amylase increased (Investigations) | 0 | 1 | 0
Biopsy lymph gland (Investigations) | 1 | 0 | 0
Oxygen saturation decreased (Investigations) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Seronegative arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Anal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Enchondromatosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Retinal melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Spinal cord neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Carotid artery aneurysm (Nervous system disorders) | 1 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 2 | 0 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 0
Essential tremor (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 3 | 0 | 0
Hemiparesis (Nervous system disorders) | 1 | 0 | 0
Loss of consciousness (Nervous system disorders) | 2 | 0 | 0
Paraparesis (Nervous system disorders) | 1 | 0 | 0
Radiculopathy (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
Device breakage (Product Issues) | 0 | 1 | 0
Device loosening (Product Issues) | 1 | 0 | 0
Adjustment disorder (Psychiatric disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Completed suicide (Psychiatric disorders) | 1 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 3
Drug abuse (Psychiatric disorders) | 2 | 0 | 0
Major depression (Psychiatric disorders) | 0 | 1 | 1
Personality disorder (Psychiatric disorders) | 1 | 0 | 0
Schizophrenia (Psychiatric disorders) | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 1 | 3
Suicide attempt (Psychiatric disorders) | 2 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 3 | 1 | 1
Bladder mass (Renal and urinary disorders) | 0 | 1 | 0
Calculus urinary (Renal and urinary disorders) | 1 | 0 | 0
Renal colic (Renal and urinary disorders) | 1 | 0 | 0
Cystocele (Reproductive system and breast disorders) | 1 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Bereavement (Social circumstances) | 0 | 0 | 1
Aortic stenosis (Vascular disorders) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 0 | 1
Lymphocele (Vascular disorders) | 1 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 1
Peripheral artery stenosis (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | D/C/F/TAF (Test) (Baseline to End of Extension [EOE]) (N=763) | Control (Baseline to Switch) (N=378) | Switch to D/C/F/TAF Group (N=352)
Abdominal pain (Gastrointestinal disorders) | 64 | 7 | 9
Diarrhoea (Gastrointestinal disorders) | 104 | 18 | 40
Nausea (Gastrointestinal disorders) | 41 | 8 | 12
Vomiting (Gastrointestinal disorders) | 41 | 4 | 6
Fatigue (General disorders) | 54 | 13 | 19
Bronchitis (Infections and infestations) | 73 | 10 | 21
Gastroenteritis (Infections and infestations) | 44 | 12 | 15
Influenza (Infections and infestations) | 53 | 7 | 10
Nasopharyngitis (Infections and infestations) | 144 | 42 | 42
Pharyngitis (Infections and infestations) | 58 | 11 | 14
Sinusitis (Infections and infestations) | 52 | 12 | 13
Syphilis (Infections and infestations) | 57 | 13 | 20
Upper respiratory tract infection (Infections and infestations) | 163 | 39 | 56
Vitamin D deficiency (Metabolism and nutrition disorders) | 74 | 29 | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 84 | 9 | 22
Back pain (Musculoskeletal and connective tissue disorders) | 107 | 23 | 31
Osteopenia (Musculoskeletal and connective tissue disorders) | 49 | 22 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 51 | 15 | 14
Headache (Nervous system disorders) | 93 | 18 | 29
Depression (Psychiatric disorders) | 41 | 12 | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 75 | 17 | 21
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 43 | 13 | 7
Rash (Skin and subcutaneous tissue disorders) | 43 | 6 | 12
Hypertension (Vascular disorders) | 47 | 7 | 11

LIMITATIONS AND CAVEATS:
The limitation of the study was the open-label design.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2015-05-29): https://cdn.clinicaltrials.gov/large-docs/17/NCT02269917/Prot_002.pdf
  • Statistical Analysis Plan (2018-03-28): https://cdn.clinicaltrials.gov/large-docs/17/NCT02269917/SAP_003.pdf